CLINICAL TRIAL: NCT02938533
Title: Pilot Study of a Multi-Pronged Intervention Using Social Norms and Priming to Improve Adherence to Antiretroviral Therapy and Retention in Care Among Adults Living With HIV in Tanzania
Brief Title: Social Norms and Priming to Improve Adherence to Antiretroviral Therapy and Retention in Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: Ministry of Health, Tanzania (Other Government); Mexican National Institute of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: OPP1118511
Record Dates: First submitted 2016-10-11; First posted 2016-10-19 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: HIV Infection; Adherence
MeSH Terms: conditions — HIV Infections | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (No Intervention): Standard HIV primary care services available at HIV care and treatment clinics in Tanzania.
- Behavioral Intervention Using Social Norms and Priming (Experimental): Patients in this arm may have been exposed to the behavioral intervention, which included the following components: 1) visual feedback about clinic-level retention in care through an interactive poster; 2) a self-relevant priming image that appeared on all components; and 3) a take-home item (i.e., pillbox or calendar) with the priming image.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — The intervention includes a clinic-based component and a take-home component. All components include the priming image of a Baobab tree. The clinic-based component is an interactive poster that rewarded appointment attendance. Patients who attend three consecutive on-time visits are congratulated and given a colored sticker to place on a poster that is publicly displayed at the clinic. In one clinic, the take-home component is a 2015 calendar in Kiswahili that contained the priming Baobab image. In the other clinic, the take-home component is a small plastic pillbox featuring the Baobab logo.
  Arms: Behavioral Intervention Using Social Norms and Priming

SUMMARY:
Interventions incorporating constructs from behavioral economics and psychology have the potential to enhance HIV 'treatment as prevention' (TasP) strategies. To test this hypothesis, the investigators evaluated a combination intervention to improve antiretroviral therapy (ART) adherence based on the concepts of social norms and priming.

DETAILED DESCRIPTION:
The investigators conducted a quasi-experimental pilot study of a combination behavioral intervention based on the concepts of social norms and priming. The intervention included visual feedback about clinic-level retention in care, a self-relevant prime, and useful take-home items with the priming image. The intervention was developed using tools from marketing research and patient-centered design. The hypothesis was that the intervention would improve retention in care and adherence to ART among patients living with HIV infection (PLHIV). The intervention was implemented at two HIV primary clinics in Shinyanga, Tanzania in 2-week intervals for six months. The investigators reviewed medical records of a random sample of exposed and unexposed adult PLHIV to compare retention and the proportion of patients with medication possession ratio (MPR) ≥95% after six months.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Living with HIV infection
3. Receiving HIV primary care at one of the two study clinics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2015-08; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Retention in care, defined as an attended visit between 150-210 days after the baseline visit | 6 months
  This measure of retention in care accounts for variability in visit scheduling by individual providers and therefore uses a window period of 150-210 days to determine whether the patient was in care at 6 months
>=95% medication possession ratio (MPR) | 6 months
  MPR is a measure of ART adherence that is correlated with viral suppression

SECONDARY OUTCOMES:
The proportion of scheduled visits that were completed during the 6-month observation period | 6 months
Medication possession ratio (MPR), continuous scale | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sandra I McCoy, PhD, Principal Investigator — University of California, Berkeley
Locations (2):
- Tanzania (2):
  - Bugsi Dispensary, Kahama, Shinyanga
  - Tinde Health Center, Shinyanga

REFERENCES:
- [Derived] McCoy SI, Fahey C, Rao A, Kapologwe N, Njau PF, Bautista-Arredondo S. Pilot study of a multi-pronged intervention using social norms and priming to improve adherence to antiretroviral therapy and retention in care among adults living with HIV in Tanzania. PLoS One. 2017 May 9;12(5):e0177394. doi: 10.1371/journal.pone.0177394. eCollection 2017. PMID 28486553